CLINICAL TRIAL: NCT00289471
Title: Dementia in Primary Care: Setting the Stage for Quality Improvement
Brief Title: Identifying Patients With Dementia in Primary Care
Acronym: GEMS
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: IIR 05-112
Record Dates: First submitted 2006-02-08; First posted 2006-02-09 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Dementia; Memory Disorders
Keywords: Sensitivity and specificity; Physician's practice patterns; Health Care costs; Quality of Health Care
MeSH Terms: conditions — Dementia; Memory Disorders; Hypersensitivity

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cognitive Screening: Cognitive screening
  Interventions: Other: No intervention delivered.

INTERVENTIONS:
Other: No intervention delivered. — No intervention delivered.

SUMMARY:
Veterans who completed GEMS-Phase 1 will be asked to participate in GEMS-Phase 2 to determine the accuracy of methods used to assess mild memory problems. This will better help us evaluate the screening test completed in GEMS-Phase 1. The goals are:

1. Compare the assessment of memory made at the initial visit to assessments of memory made at the second evaluation.
2. Determine of veterans with mild memory problems have improvement or worsening of these memory problems over time. Our long-term goal remains to optimize the quality of care for veterans with cognitive impairment. We will also determine if patient characteristics can be used to target case-finding, describe the current process of care and evaluate the association between cognitive impairment and overall- and dementia-related health care utilization and costs.

DETAILED DESCRIPTION:
Dementia has high public health significance due to its prevalence, adverse impact on patients and caregivers, high economic cost to society and the rapidly expanding numbers of individuals age 65 and older. As the largest provider of geriatric care in the U.S., dementia is particularly relevant to the Veterans Health Administration (VHA). However, only a small proportion of patients with dementia are diagnosed early when treatments are most effective and the opportunity for careful life planning remains, in part because of the absence of feasible, well-validated case-finding instruments. Our long-term objective is to improve the care and outcomes of veterans with clinically significant cognitive impairment. The first steps towards realizing this objective are to determine the acceptability of cognitive screening to patients and to identify feasible, valid case-finding tools for primary care. We will also determine if patient characteristics can be used to target case-finding, describe the current process of care and evaluate the association between cognitive impairment and overall- and dementia-related health care utilization and costs. Our research team, located in the Center for Health Services Research in Primary Care, brings together researchers uniquely suited to achieving this objective. Specific Aims1.Primary Aim: To determine if cognitive screening is acceptable to patients, and whether brief cognitive screeners perform as well as the longer Modified Mini-Mental Status Exam (3MS) for dementia and cognitive impairment-not dementia (CIND).Primary Hypothesis 1: Higher perceived risk of dementia, higher perceived benefits and fewer perceived harms from screening will be positively associated with screening acceptance. Primary Hypotheses 2: Compared to the 3MS, the Mini-Cog, Memory Impairment Screen and 2-item functional screen will have similar performance characteristics. 2.Secondary Aim 1: To determine if sociodemographic and clinical characteristics available in the electronic medical record can be used to target individuals for cognitive screening and improve screening accuracy. Hypothesis: The combination of sociodemographic characteristics/clinical information and screening results will more accurately discriminate between demented and non-demented patients than screening results alone.3.Secondary Aim 2: To describe current care for an inception cohort with dementia or cognitive impairment-not dementia. Hypothesis: Compared to patients with dementia, patients with cognitive impairment-not dementia will undergo less diagnostic testing, be less likely to complete an advanced directive and be less likely to receive dementia specific medications. 4.Exploratory Aim: To evaluate the association between cognitive impairment and overall- and dementia-related health care utilization and costs. Exploratory Hypothesis: Controlling for sociodemographic characteristics and medical comorbidity, overall healthcare utilization and costs will increase as cognitive impairment increases. In phase 1, a random sample of primary care patients age 65 years will be recruited from 3 primary care clinics to complete the Modified Dementia Screening Acceptance and Perceived Harms Questionnaire. In phase 2, patients will complete three brief instruments and the standard 15-item 3MS that will be compared to a criterion standard interview for dementia. We project 140-200 patients will have dementia, 200-300 CIND, and approximately 600 will be cognitively normal. Instruments will be compared using sensitivity/specificity, likelihood ratios and receiver operating characteristic curves. The emotional impact of screening will be assessed following screening. Clinical and sociodemographic characteristics available in the Computerized Patient Record System, together with cognitive screening results, will be analyzed with logistic regression models to identify risk factors that may be used to target individuals for cognitive screening and/or improve screening accuracy. Care patterns for patients with dementia and CIND will be described based on detailed chart abstractions. For the exploratory analysis on cognitive impairment and utilization, two-part utilization models will be estimated for each utilization type, outpatient clinic visits, inpatient visits, pharmacy utilization, and other utilization types; utilization data will be obtained from administrative data.

ELIGIBILITY:
Inclusion Criteria:

* Previous participant who completed GEMS-Phase 1
* Continues to be a VA clinic patient
* Identifies a key informant with phone

Exclusion Criteria:

* Severe hearing or visual impairment
* Acute medical condition

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Veterans' who have previously completed GEMS-Phase 1 testing, continues to be a VA clinic patient and identifies a key family member or friend who will answer questions about the veteran's memory and daily activities.
Sampling Method: Probability Sample
Enrollment: 630 (Actual)
Dates: Start 2009-10; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John W Williams, MD MHS, Principal Investigator — Durham VA Medical Center
Locations (1):
- Durham VA Medical Center HSR&D COE, Durham, North Carolina, United States

REFERENCES:
- [Result] Plassman BL, Williams JW Jr, Burke JR, Holsinger T, Benjamin S. Systematic review: factors associated with risk for and possible prevention of cognitive decline in later life. Ann Intern Med. 2010 Aug 3;153(3):182-93. doi: 10.7326/0003-4819-153-3-201008030-00258. Epub 2010 Jun 14. PMID 20547887
- [Result] Holsinger T, Plassman BL, Stechuchak KM, Burke JR, Coffman CJ, Williams JW Jr. Screening for cognitive impairment: comparing the performance of four instruments in primary care. J Am Geriatr Soc. 2012 Jun;60(6):1027-36. doi: 10.1111/j.1532-5415.2012.03967.x. Epub 2012 May 30. PMID 22646750

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cognitive Screening
Started | 630
Completed | 630
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cognitive Screening
Number analyzed (Participants) | 630
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.8 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 585
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 165
  White | 461
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 630

OUTCOME MEASURES:

1. Primary Outcome: Performance Characteristics
Description: Sensitivity and Specificity for Modified Mini-Mental Status Examination (MMSE), a measure scored 0-100 to assess cognitive impairment
Time Frame: Cross-sectional [at baseline; no longitudinal component]
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cognitive Screening
Number analyzed (Participants) | 630
Percentage of participants
  Sensitivity (%) | 86 [64 to 95]
  Specificity (%) | 79 [72 to 82]

ADVERSE EVENTS:
Time Frame: Cross-sectional [at baseline; no longitudinal component]
Arm/Group | Cognitive Screening
Serious Adverse Events (participants affected / at risk) | 0/630
Other Adverse Events (participants affected / at risk) | 0/630

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes